CLINICAL TRIAL: NCT02156414
Title: Lymph Node Involvement Using Extended Pelvic Lymphadenectomy in Clinically Localized Prostate Cancer in Bogota Colombia.
Brief Title: Lymph Node Involvement Using Extended Pelvic Lymphadenectomy in Clinically Localized Prostate Cancer
Acronym: LNIEPLCLPC
Status: Completed | Type: Observational
Sponsor: Javeriana University (Other)
Collaborators: Hospital Universitario San Ignacio (Other); Fundación Santa Fe de Bogota (Other); Fundación Cardioinfantil Instituto de Cardiología (Other)
Responsible Party: Principal Investigator, Jose Gustavo Ramos, MD, Urology Resident, Javeriana University
Other Study IDs: 7-2013
Record Dates: First submitted 2014-05-13; First posted 2014-06-05 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Secondary Malignant Neoplasm of Lymph Node; Prostatic Neoplasms
Keywords: Prostatectomy; Extended Lymphadenectomy; Pelvic lymph node dissection; Prostatic Neoplasm; Prospective Studies
MeSH Terms: conditions — Lymphatic Metastasis; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clinically Localized Prostatic Neoplasm: Radical Prostatectomy Extended Lymphadenectomy
  Interventions: Procedure: Radical Prostatectomy; Procedure: Extended Lymphadenectomy

INTERVENTIONS:
Procedure: Radical Prostatectomy — Radical Prostatectomy
Procedure: Extended Lymphadenectomy — Extended Lymphadenectomy

SUMMARY:
Prostate cancer is considered the fourth most common malignancy cancer in America. However, in Colombia the incidence is higher, and it is considered the second cause of death among men for malignance diseases. In the framework of clinical localized prostate cancer there is a controversy regarding the best predictors of risk and the best treatment options. The actual literature is discussing the possibility of underestimate the disease and actual tools are not sufficient for proper characterization. Is in this context that extended pelvic lymphadenectomy emerges as a stratification tool in prostate cancer that defines the real commitment of the disease. The investigators need to know the characteristics that the disease has on the investigators community so the investigators can generate appropriate therapeutic approach. Thus, the present prospective observational-descriptive multicenter study, want to determine in three referral centers in Bogotá Colombia , the frequency of pelvic node involvement in patients with localized clinical prostate cancer from the stratification achieved by pelvic lymphadenectomy extended.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical localized prostate cancer
* Clinical stage: cT1-cT2-, N0-Nx, M0-Mx
* Patients who undergo radical prostatectomy and extended lymphadenectomy in one of the 3 centers of reference.

Exclusion Criteria:

* Patients in which the standard technique of the extended lymphadenectomy could not be done and it was changed.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical localized prostate cancer who undergo a radical prostatectomy in the 3 centers. Hospital Universitario San Ignacio, Hospital Fundacion Santa fe de Bogota, Fundacion Cardioinfantil.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Lymph Node Involvement Using Extended Pelvic Lymphadenectomy by histopathology analysis | within the first 30 days after surgery
  After extended pelvic lymphadenectomy the nodes are classified in ilio-obturator nodes and internal iliaca nodes. Then those nodes are send to the pathology department of the each center, and by the histopathology analysis, the pathologist determine which nodes are compromised. With the histopathology result, the investigators report de nodal involvement.

SECONDARY OUTCOMES:
The Histopathology substaging Gleason score in the surgery piece vs Biopsy report before surgery. | Within the first 30 days after surgery
  After radical prostatectomy the specimen (prostate) is send to the pathology department of each center, and by the histopathology analysis, the pathologist determine the gleason score. Then the investigators compare this result to the one achieved in the biopsy result, and determine if there was a oncologic substaging related to the gleason score.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE G RAMOS, MF, Principal Investigator — Javeriana University; JUAN G CATAÑO, MD, Study Director — Javeriana University; LUIS G VILLARRAGA, MD, Study Chair — Javeriana University
Locations (3):
- Colombia (3):
  - Fundacion Cardioinfantil, Bogotá, Bogota D.C.
  - Fundacion Hospital Santafe, Bogotá, Bogota D.C.
  - Hospital Universitario San Ignacio, Bogotá, Bogota D.C.

REFERENCES:
- [Background] Heidenreich A, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Mottet N, Schmid HP, van der Kwast T, Wiegel T, Zattoni F. [EAU guidelines on prostate cancer. Part I: screening, diagnosis, and treatment of clinically localised disease]. Actas Urol Esp. 2011 Oct;35(9):501-14. doi: 10.1016/j.acuro.2011.04.004. Epub 2011 Jul 14. Spanish. PMID 21757259
- [Background] Delahunt B, Miller RJ, Srigley JR, Evans AJ, Samaratunga H. Gleason grading: past, present and future. Histopathology. 2012 Jan;60(1):75-86. doi: 10.1111/j.1365-2559.2011.04003.x. PMID 22212079
- [Background] Briganti A, Chun FK, Salonia A, Gallina A, Zanni G, Scattoni V, Valiquette L, Rigatti P, Montorsi F, Karakiewicz PI. Critical assessment of ideal nodal yield at pelvic lymphadenectomy to accurately diagnose prostate cancer nodal metastasis in patients undergoing radical retropubic prostatectomy. Urology. 2007 Jan;69(1):147-51. doi: 10.1016/j.urology.2006.09.008. PMID 17270638
- [Background] Abdollah F, Sun M, Suardi N, Gallina A, Capitanio U, Bianchi M, Tutolo M, Passoni N, Karakiewicz PI, Rigatti P, Montorsi F, Briganti A; National Comprehensive Cancer Network. National Comprehensive Cancer Network practice guidelines 2011: Need for more accurate recommendations for pelvic lymph node dissection in prostate cancer. J Urol. 2012 Aug;188(2):423-8. doi: 10.1016/j.juro.2012.03.129. Epub 2012 Jun 13. PMID 22698627
- [Background] Abdollah F, Sun M, Briganti A, Thuret R, Schmitges J, Gallina A, Suardi N, Capitanio U, Salonia A, Shariat SF, Perrotte P, Rigatti P, Montorsi F, Karakiewicz PI. Critical assessment of the European Association of Urology guideline indications for pelvic lymph node dissection at radical prostatectomy. BJU Int. 2011 Dec;108(11):1769-75. doi: 10.1111/j.1464-410X.2011.10204.x. Epub 2011 Apr 20. PMID 21507189
- [Background] Mohler J, Bahnson RR, Boston B, Busby JE, D'Amico A, Eastham JA, Enke CA, George D, Horwitz EM, Huben RP, Kantoff P, Kawachi M, Kuettel M, Lange PH, Macvicar G, Plimack ER, Pow-Sang JM, Roach M 3rd, Rohren E, Roth BJ, Shrieve DC, Smith MR, Srinivas S, Twardowski P, Walsh PC. NCCN clinical practice guidelines in oncology: prostate cancer. J Natl Compr Canc Netw. 2010 Feb;8(2):162-200. doi: 10.6004/jnccn.2010.0012. No abstract available. PMID 20141676
- [Background] Thompson I, Thrasher JB, Aus G, Burnett AL, Canby-Hagino ED, Cookson MS, D'Amico AV, Dmochowski RR, Eton DT, Forman JD, Goldenberg SL, Hernandez J, Higano CS, Kraus SR, Moul JW, Tangen CM; AUA Prostate Cancer Clinical Guideline Update Panel. Guideline for the management of clinically localized prostate cancer: 2007 update. J Urol. 2007 Jun;177(6):2106-31. doi: 10.1016/j.juro.2007.03.003. No abstract available. PMID 17509297
- [Background] Gacci M, Del Popolo G, Artibani W, Tubaro A, Palli D, Vittori G, Lapini A, Serni S, Carini M. Visual assessment of uroflowmetry curves: description and interpretation by urodynamists. World J Urol. 2007 Jun;25(3):333-7. doi: 10.1007/s00345-007-0165-8. Epub 2007 Apr 14. PMID 17436003
- [Background] Boyle P, Ferlay J. Cancer incidence and mortality in Europe, 2004. Ann Oncol. 2005 Mar;16(3):481-8. doi: 10.1093/annonc/mdi098. Epub 2005 Feb 17. PMID 15718248
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for prostate cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Jul 17;157(2):120-34. doi: 10.7326/0003-4819-157-2-201207170-00459. PMID 22801674
- [Background] Miki J, Egawa S. The role of lymph node dissection in the management of prostate cancer. Int J Clin Oncol. 2011 Jun;16(3):195-202. doi: 10.1007/s10147-011-0245-z. Epub 2011 May 10. PMID 21556799
- [Background] Wagner M, Sokoloff M, Daneshmand S. The role of pelvic lymphadenectomy for prostate cancer--therapeutic? J Urol. 2008 Feb;179(2):408-13. doi: 10.1016/j.juro.2007.09.027. PMID 18076938
- [Background] Epstein JI, Allsbrook WC Jr, Amin MB, Egevad LL; ISUP Grading Committee. The 2005 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma. Am J Surg Pathol. 2005 Sep;29(9):1228-42. doi: 10.1097/01.pas.0000173646.99337.b1. No abstract available. PMID 16096414
- [Background] Harnden P, Shelley MD, Coles B, Staffurth J, Mason MD. Should the Gleason grading system for prostate cancer be modified to account for high-grade tertiary components? A systematic review and meta-analysis. Lancet Oncol. 2007 May;8(5):411-9. doi: 10.1016/S1470-2045(07)70136-5. PMID 17466898
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] D'Amico AV, Cote K, Loffredo M, Renshaw AA, Schultz D. Determinants of prostate cancer-specific survival after radiation therapy for patients with clinically localized prostate cancer. J Clin Oncol. 2002 Dec 1;20(23):4567-73. doi: 10.1200/JCO.2002.03.061. PMID 12454114
- [Background] Allaf ME, Palapattu GS, Trock BJ, Carter HB, Walsh PC. Anatomical extent of lymph node dissection: impact on men with clinically localized prostate cancer. J Urol. 2004 Nov;172(5 Pt 1):1840-4. doi: 10.1097/01.ju.0000140912.45821.1d. PMID 15540734
- [Background] Bader P, Burkhard FC, Markwalder R, Studer UE. Disease progression and survival of patients with positive lymph nodes after radical prostatectomy. Is there a chance of cure? J Urol. 2003 Mar;169(3):849-54. doi: 10.1097/01.ju.0000049032.38743.c7. PMID 12576797
- [Background] Clark T, Parekh DJ, Cookson MS, Chang SS, Smith ER Jr, Wells N, Smith J Jr. Randomized prospective evaluation of extended versus limited lymph node dissection in patients with clinically localized prostate cancer. J Urol. 2003 Jan;169(1):145-7; discussion 147-8. doi: 10.1016/S0022-5347(05)64055-4. PMID 12478123
- [Background] Briganti A, Blute ML, Eastham JH, Graefen M, Heidenreich A, Karnes JR, Montorsi F, Studer UE. Pelvic lymph node dissection in prostate cancer. Eur Urol. 2009 Jun;55(6):1251-65. doi: 10.1016/j.eururo.2009.03.012. Epub 2009 Mar 10. PMID 19297079
- [Background] Heidenreich A, Bellmunt J, Bolla M, Joniau S, Mason M, Matveev V, Mottet N, Schmid HP, van der Kwast T, Wiegel T, Zattoni F; European Association of Urology. EAU guidelines on prostate cancer. Part 1: screening, diagnosis, and treatment of clinically localised disease. Eur Urol. 2011 Jan;59(1):61-71. doi: 10.1016/j.eururo.2010.10.039. Epub 2010 Oct 28. PMID 21056534
- [Background] Cagiannos I, Karakiewicz P, Eastham JA, Ohori M, Rabbani F, Gerigk C, Reuter V, Graefen M, Hammerer PG, Erbersdobler A, Huland H, Kupelian P, Klein E, Quinn DI, Henshall SM, Grygiel JJ, Sutherland RL, Stricker PD, Morash CG, Scardino PT, Kattan MW. A preoperative nomogram identifying decreased risk of positive pelvic lymph nodes in patients with prostate cancer. J Urol. 2003 Nov;170(5):1798-803. doi: 10.1097/01.ju.0000091805.98960.13. PMID 14532779
- [Background] Abdollah F, Sun M, Thuret R, Budaus L, Jeldres C, Graefen M, Briganti A, Perrotte P, Rigatti P, Montorsi F, Karakiewicz PI. Decreasing rate and extent of lymph node staging in patients undergoing radical prostatectomy may undermine the rate of diagnosis of lymph node metastases in prostate cancer. Eur Urol. 2010 Dec;58(6):882-92. doi: 10.1016/j.eururo.2010.09.029. Epub 2010 Sep 28. PMID 20932637
- [Background] Bhatta-Dhar N, Reuther AM, Zippe C, Klein EA. No difference in six-year biochemical failure rates with or without pelvic lymph node dissection during radical prostatectomy in low-risk patients with localized prostate cancer. Urology. 2004 Mar;63(3):528-31. doi: 10.1016/j.urology.2003.09.064. PMID 15028451
- [Background] Hyndman ME, Mullins JK, Pavlovich CP. Pelvic node dissection in prostate cancer: extended, limited, or not at all? Curr Opin Urol. 2010 May;20(3):211-7. doi: 10.1097/MOU.0b013e328338405d. PMID 20224412
- [Background] Gerstenbluth RE, Seftel AD, Hampel N, Oefelein MG, Resnick MI. The accuracy of the increased prostate specific antigen level (greater than or equal to 20 ng./ml.) in predicting prostate cancer: is biopsy always required? J Urol. 2002 Nov;168(5):1990-3. doi: 10.1016/S0022-5347(05)64279-6. PMID 12394692
- [Result] Brawley OW. Prostate cancer epidemiology in the United States. World J Urol. 2012 Apr;30(2):195-200. doi: 10.1007/s00345-012-0824-2. Epub 2012 Apr 5. PMID 22476558